CLINICAL TRIAL: NCT03318536
Title: Effect of Granisetron on Usage of Sympathomimetics During Caesarean Section - a Retrospective Analysis
Brief Title: Effect of Granisetron on Usage of Sympathomimetics During Caesarean Section
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Florian Raimann, Dr. med. Florian Raimann, Johann Wolfgang Goethe University Hospital
Other Study IDs: XXX/17
Record Dates: First submitted 2017-10-09; First posted 2017-10-24 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Hypotension; Cesarean Section Complications
Keywords: Serotonin Antagonists; Sympathomimetics
MeSH Terms: conditions — Hypotension | interventions — Granisetron

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- No Granisetron: 120 Patients prior to changes of intern standards of caesarean section. Before march 2017 no patient undergoing elective caesarean section received Granisetron as a matter of routine.
  Interventions: Drug: No Granisetron
- With Granisetron: 120 Patients after changes of intern standards of caesarean section. After march 2017 all patient undergoing elective caesarean section received Granisetron as a matter of routine.
  Interventions: Drug: Granisetron Hydrochloride

INTERVENTIONS:
Drug: Granisetron Hydrochloride — Patients received Granisetron.
  Other Names: Granisetron; 5-hydroxytryptamine 3 receptor antagonist
  Groups: With Granisetron
Drug: No Granisetron — Patients who did not receive Granisetron.
  Groups: No Granisetron

SUMMARY:
The aim of the present study is to quantify the dose and usage of sympathomimetics used in caesarean section.

DETAILED DESCRIPTION:
Recent metaanalysis showed significantly reduced hypotension and bradycardia in patients undergoing caesarean section in spinal anesthesia when 5-hydroxytryptamine 3 receptor antagonists were used prophylactically.

Due to this fact in our clinic the standard procedure was changed. All patients for caesarean section receive Granisetron before spinal anesthesia.

The aim of the present study is to evaluate the usage and dose of sympathomimetics during spinal anesthesia.

Therefore the investigators will evaluate approximately 120 participants who received granisetron and 120 participants who did not receive 5-hydroxytryptamine 3 receptor antagonists.

ELIGIBILITY:
Inclusion Criteria:

* caesarean section in spinal anesthesia

Exclusion Criteria:

* withdrawal
* incomplete documentation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients who underwent spinal anesthesia for caesarean section in out clinic.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Sympathomimetics | 30 minutes starting with induction of spinal anesthesia.
  Type of sympathomimetics during during the operation

SECONDARY OUTCOMES:
Sympathomimetics | 30 minutes starting with induction of spinal anesthesia.
  Cumulative dose of sympathomimetics during during the operation
Volume substitution | 30 minutes starting with induction of spinal anesthesia.
  Type of perioperative infused volume during the operation
Volume substitution | 30 minutes starting with induction of spinal anesthesia.
  Cumulative volume of perioperative infused volume during the operation
Haemotherapy | 30 minutes starting with induction of spinal anesthesia.
  Type of haemotherapy.
Haemotherapy | 30 minutes starting with induction of spinal anesthesia.
  Cumulative volume of haemotherapy.
Duration until first application of sympathomimetics | 30 minutes starting with induction of spinal anesthesia.
  Duration until first administration of any kind of sympathomimetics.
Oxytocin | 30 minutes starting with induction of spinal anesthesia.
  Duration until first administration of oxytocin.
Oxytocin | 30 minutes starting with induction of spinal anesthesia.
  Cumulative dose of Oxytocin.
Uterotonic agents | 30 minutes starting with induction of spinal anesthesia.
  Kind of uterotonic agents.
Uterotonic agents | 30 minutes starting with induction of spinal anesthesia.
  Cumulative dose of uterotonic agents.

CONTACTS AND LOCATIONS:
Overall Officials: Kai Zacharowski, Prof. Dr. med., Study Director — Department of Anesthesia, Intensive Care Medicine and Pain Therapy
Locations (1):
- Klinikum Goethe Universität Frankfurt am Main, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raimann FJ, Baldauf HP, Louwen F, Jennewein L, Fischer D, Zacharowski K, Weber CF. Granisetron reduces the need for uterotonics but not sympathomimetics during cesarean delivery. Int J Gynaecol Obstet. 2019 Jun;145(3):361-366. doi: 10.1002/ijgo.12819. Epub 2019 Apr 15. PMID 30932170